CLINICAL TRIAL: NCT04405765
Title: Prospective, Randomized, Single-Center Study to Compare Clinical Outcomes Between Cryopreserved and Lyopreserved Stravix as an Adjunct to NPWT in the Treatment of Complex Wounds
Brief Title: Cryopreserved vs. Lyopreserved Stravix as an Adjunct to NPWT in the Treatment of Complex Wounds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Osiris Therapeutics (Industry)
Responsible Party: Principal Investigator, Larry Lavery, Professor and Director of Research, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0293
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Wound
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, 2-arm parallel assignment, randomized clinical trial. Stravix will be applied at initial visit with NPWT and will only be reapplied after 4 weeks if wound is not ready for grafting unless debridement is indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Lyopreserved Stravix (Active Comparator): Treated with NPWT and lyopreserved Stravix
  Interventions: Device: NPWT and lyopreserved Stravix
- Cryopreserved Stravix (Active Comparator): Treated with NPWT and cryopreserved Stravix
  Interventions: Device: NPWT and cryopreserved Stravix

INTERVENTIONS:
Device: NPWT and lyopreserved Stravix — Subjects will be treated with NPWT and lyopreserved Stravix
  Arms: Lyopreserved Stravix
Device: NPWT and cryopreserved Stravix — Subjects will be treated with NPWT and lyopreserved Stravix
  Arms: Cryopreserved Stravix

SUMMARY:
This study is a prospective, 2-arm parallel assignment, randomized clinical trial to compare lyopreserved vs cryopreserved Stravix as an adjunct therapy to NPWT.

DETAILED DESCRIPTION:
Screening

1. Explain purpose and nature of the study and obtain signature on the informed consent document.

2. Screen the subject against protocol inclusion and exclusion criteria, including all pertinent tests, including pregnancy test 3. Complete SF-36, EuroQol 5 dimensions (EQ-5D) and PROMIS® Baseline (may be done as same day as screening procedures or within +2 days of screening and before start of Therapy/Treatment Phase)

1. Obtain general medical history and demographic information and social history
2. Complete a physical examination, body weight, height, and vital signs, including measurement of resting heart rate, respiratory rate, and blood pressure while seated.
3. Select target study ulcer
4. Obtain complete history pertinent to DFU disease including duration of the target ulcer, previous and current treatment. Document ulcer classification.
5. Perform debridement and obtain tissue collection (3 tissue and 1 bone).
6. Perform standardized photography and measurement of the study wound (eKare or available camera with ruler). Assess the post-debridement ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device (eKare, Fairfax, VA). These values are the baseline measurements for calculating wound closure rate at the two-week run-in visit.
7. Perform hyperspectral imaging of dorsal and plantar aspects of the foot.
8. Perform neuropathy assessment
9. Collect all relevant concomitant medication (antibiotics, antifungals and other anti-infective therapies)
10. Place Stravix (lyo or cryo per randomization schedule) and dress wound for NPWT therapy.
11. Document size of Stravix used.
12. Disburse subject stipend Therapy/Treatment Phase (Weekly visits +/- 4 days)

Study Visit 1-11:

1. Assess target ulcer (if wound has closed, document as such, skip to step 5).
2. Document time on/off NPWT if applicable.
3. Perform standardized photography of the study wound when NPWT is removed.
4. If Stravix is removed, assess the ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device - if the wound is deemed closed by the physician, skip to EOS visit.
5. Perform hyperspectral imaging of the dorsal and plantar aspects of the foot if wound is active or closed.
6. Debride wound if indicated. Re-measure wound if surgical debridement is performed prior to dressing the wound.
7. Collect all relevant concomitant medication.
8. If wound is still active, redress the wound with assigned Stravix (if removed for debridement) and NPWT. Document all dressings applied including size of Stravix.
9. Disburse subject stipend
10. Note: at week 4, if wound is not ready for grafting, remove existing Stravix and replace with new piece of Stravix (per randomization schedule)
11. Assess for AE/SAEs and/or follow up on previous AE/SAEs.

Study Visit Closed 1. When a subject's study wound has closed, they will perform the EOS evaluation.

Study Visit 12/EOS:

1. At the time of wound closure, subjects will perform EOS visit.
2. A subject whose wound is not deemed closed (epithelialized with no drainage) by physician at week 12 will exit from the study after the week 12 wound evaluation.
3. Assess index ulcer.
4. If wound has not closed, perform standardized photography of the study wound.
5. If wound has not closed, assess the ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device.
6. Perform hyperspectral imaging of the dorsal and plantar aspects of the foot if wound is active or healed.
7. If wound has not closed, redress the wound per physician-directed standard of care.
8. Administer Patient Reported Outcome (PRO) (questionnaires).
9. Collect all relevant concomitant medication
10. Perform EOS visit documentation
11. Follow up on AE/SAEs that have been reported that have not yet been resolved.

Study Visit Follow-up:

1. If the wound heals during the treatment phase or if the wound is not healed after 12 weeks, data from their electronic medical record will be evaluated to identify healing, time to heal, adverse events related to the wound.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a diabetes mellitus
* Men/women ≥21 years old
* Post-operative foot or ankle wounds sized >4cm2 that have presented for <1 year
* ABI ≥0.5 or toe pressures >30 mmHg
* Wounds indicated for treatment with NPWT

Exclusion Criteria:

* Active Charcot arthropy
* Unable to use NPWT at home
* Untreated bone or soft tissue infection
* Is pregnant or plans to become pregnant
* Is nursing or actively lactating
* Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including untreated schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years.
* Active alcohol or substance abuse in the opinion of the investigator that could impair the subject's ability to provide informed consent, participate in the study protocol or record study materials

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lyopreserved Stravix | Cryopreserved Stravix
Started | 22 | 20
Completed | 21 | 19
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lyopreserved Stravix | Cryopreserved Stravix | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (11.5) | 55.4 (6.4) | 52.85 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 17 | 16 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5 | 1 | 6
  African American | 6 | 5 | 11
  Hispanic | 10 | 9 | 19
  Other | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Wound Closure
Description: Number of patients who achieve wound closure (complete epithelialization with no drainage)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lyopreserved Stravix | Cryopreserved Stravix
Number analyzed (Participants) | 21 | 19
Participants | 4 | 7

2. Secondary Outcome: Duration of Negative Pressure Wound Therapy
Description: Number of days patient received negative pressure wound therapy after application of Stravix
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lyopreserved Stravix | Cryopreserved Stravix
Number analyzed (Participants) | 21 | 19
days | 8.88 (5.96) | 4.66 (2.73)

3. Secondary Outcome: Split Thickness Skin Grafting
Description: Number of patients who received a split thickness skin graft
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lyopreserved Stravix | Cryopreserved Stravix
Number analyzed (Participants) | 21 | 19
Participants | 2 | 3

4. Secondary Outcome: Infection
Description: Number of patients who developed infection
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lyopreserved Stravix | Cryopreserved Stravix
Number analyzed (Participants) | 21 | 19
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Lyopreserved Stravix | Cryopreserved Stravix
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/19
Serious Adverse Events (participants affected / at risk) | 3/21 | 2/19
Other Adverse Events (participants affected / at risk) | 1/21 | 2/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyopreserved Stravix (N=21) | Cryopreserved Stravix (N=19)
Hospital admission for foot infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospital admission for non-foot reason (General disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyopreserved Stravix (N=21) | Cryopreserved Stravix (N=19)
Infection of study wound (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT04405765/Prot_SAP_000.pdf